CLINICAL TRIAL: NCT06881082
Title: Cross-section Band Ligation Versus Stepladder Band Ligation Techniques in Prophylaxis of Esophageal Varices in Cirrhotic Liver Disease. A Randomized Controlled Trial.
Brief Title: Cross-section Band Ligation Versus Stepladder Band Ligation of Esophageal Varices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Lecturer of Tropical Medicine, Tanta University
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR978/12/24
Record Dates: First submitted 2025-03-04; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Varices
Keywords: Band ligation; esophageal varices prophylaxis
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cross-section band ligation (Experimental): 160 cirrhotic patients with endoscopic evidence of medium/large-sized esophageal varices undergoing endoscopic prophylaxis using the cross-section band ligation technique.
  Interventions: Procedure: endoscopic band ligation with cross-section technique
- stepladder band ligation (Active Comparator): 160 cirrhotic patients with endoscopic evidence of medium/large-sized esophageal varices undergoing endoscopic prophylaxis using the step ladder band ligation technique.
  Interventions: Procedure: Endoscopic band ligation using stepladder technique

INTERVENTIONS:
Procedure: endoscopic band ligation with cross-section technique — Endoscopic band ligation (EBL) of medium/large-sized esophageal varices using the cross-section banding technique. EBL will be repeated every two to four weeks until eradication. After eradication of varices, endoscopy will be repeated after 3- 6 months to check for variceal recurrence, evaluation of treatment-related side effects, bleeding rates, and mortality from EBL treatment.
  Arms: cross-section band ligation
Procedure: Endoscopic band ligation using stepladder technique — Endoscopic band ligation (EBL) of medium/large-sized esophageal varices using the stepladder banding technique. EBL will be repeated every two to four weeks until eradication. After eradication of varices, endoscopy will be repeated after 3- 6 months to check for variceal recurrence, evaluation of treatment-related side effects, bleeding rates, and mortality from EBL treatment
  Arms: stepladder band ligation

SUMMARY:
The goal of this randomized controlled trial is to evaluate the cross-section band ligation technique versus the stepladder band ligation technique in esophageal varices prophylaxis.

Researchers will compare cross-section and step ladder band ligation techniques for esophageal varices prophylaxis regarding efficacy, side effects, variceal recurrence, and survival.

Participants will undergo history-taking, clinical examination, laboratory investigations, and upper endoscopy. Index upper endoscopy will be performed to evaluate the presence, size, and grade of esophageal varices. Patients will be randomly assigned to endoscopic band ligation (EBL) either by cross-section or stepladder techniques every two to four weeks until eradication. After eradication of varices, endoscopy will be repeated after 3-6 months to check for variceal recurrence. For a period of 6 months, all patients in the treatment groups will be followed up every 3 months with clinic visits, including laboratory testing, evaluation of treatment-related side effects, bleeding rates, and mortality from EBL treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years.
* Cirrhotic patients.
* Endoscopic evidence of medium/large-sized esophageal varices.

Exclusion Criteria:

* History of variceal bleeding or previous primary prevention of varices.
* Portal vein thrombosis or previous porto-systemic shunts as TIPS.
* Patients on drugs affecting portal pressure (beta blockers, nitrates).
* Advanced cardiovascular disease including acute myocardial infarction, atrio-ventricular block, congestive heart failure, chronic peripheral ischemia, and severe bradycardia.
* Patients with severe respiratory diseases (COPD, bronchial asthma).
* Uncontrolled diabetes mellitus.
* Renal impairment.
* Hepatocellular carcinoma.
* Allergy to carvedilol.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Vriceal bleeding rate at 6 weeks follow up | through study completion, an average of 1 year
  -The occurrence of first variceal bleeding (early bleeding within 3 - 10 days after band ligation and late bleeding after that) will be evaluated and compared across the studied groups.
Mortality rate at 6 weeks follow up | through study completion, an average of 1 year
  Bleeding-related mortality rate and overall mortality rate at 6 weeks will be assessed and compared across the studied groups.
Banding side effects at 6 weeks follow up | through study completion, an average of 1 year
  Side effects of banding (e.g. post banding ulcers, portal hypertensive gastropathy, esophageal strictures and perforation) at 6 weeks will be evaluated and compared across the studied groups.

SECONDARY OUTCOMES:
Variceal obliteration rate at 6 months follow up | through study completion, an average of 1 year
  Obliteration of esophageal varices rate at 6 months will be evaluated and compared across the studied groups.
Variceal recurrence rate at 6 months follow up | through study completion, an average of 1 year
  Recurrence of esophageal varices rate at 6 months after obliteration will be evaluated and compared across the studied groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nabila A Elgazzar, MD, Principal Investigator — Tropical medicine and infectious diseases Department, Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt